CLINICAL TRIAL: NCT04020575
Title: Adoptive Immunotherapy for Advanced MUC1* Positive Breast Cancer With Autologous T Cells Engineered to Express a Chimeric Antigen Receptor, huMNC2-CAR44 or huMNC2-CAR22, Specific for a Cleaved Form of MUC1 (MUC1*)
Brief Title: Autologous huMNC2-CAR44 or huMNC2-CAR22 T Cells for Breast Cancer Targeting Cleaved Form of MUC1 (MUC1*)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minerva Biotechnologies Corporation (Industry)
Collaborators: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10038
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): Dose escalation or de-escalation is tested in cohorts of 3 patients each using standard "3+3" dose-finding.
  Interventions: Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells
- Luminal (Experimental): Dose Expansion - 15 patients will be enrolled with luminal (hormone receptor positive, HER2 negative) metastatic breast cancer.
  Interventions: Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells @ RP2D
- HER2+ (Experimental): Dose Expansion - 15 patients will be enrolled with HER2+ metastatic breast cancer.
  Interventions: Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells @ RP2D
- Triple Negative (Experimental): Dose Expansion - 15 patients will be enrolled with triple negative metastatic breast cancer.
  Interventions: Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells @ RP2D

INTERVENTIONS:
Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells — huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells are an autologous T cell product transduced with a proprietary lentiviral vector backbone coding for humanized MNC2-scFv (the targeting head).
  Arms: Dose Escalation
Biological: huMNC2-CAR44 CAR T cells or huMNC2-CAR22 CAR T cells @ RP2D — huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells are an autologous T cell product transduced with a proprietary lentiviral vector backbone coding for humanized MNC2-scFv (the targeting head) @ RP2D
  Arms: HER2+; Luminal; Triple Negative

SUMMARY:
Phase I/II study of adoptive immunotherapy for advanced MUC1* positive breast cancer with autologous T cells engineered to express either a chimeric antigen receptor, huMNC2-CAR44 or huMNC2-CAR22, which are specific for a cleaved form of MUC1 (MUC1*).

DETAILED DESCRIPTION:
Recent trials have demonstrated that chimeric antigen receptor (CAR)-modified T cells (CAR-T cells) specific for the CD19 molecule can mediate marked tumor regression in a subset of patients with advanced acute lymphoblastic leukemia (ALL) and non-Hodgkin's lymphoma (NHL). It would be ideal to extend CAR-T cell therapy to common epithelial cancers. However, this poses several challenges, including the identification of molecules expressed on tumor cells that can be targeted safely with CAR-T cells. Minerva Biotechnologies has developed a CAR T product (huMNC2-CAR44 or huMNC2-CAR22) that targets the extra cellular domain of the cleaved form of MUC1 (called MUC1*), which is the form of MUC1 that functions as a growth factor receptor and is present on large percentage of solid tumors, including breast tumors. The antibody targeting head of huMNC2-CAR44 or huMNC2-CAR22 specifically recognizes a cancerous form of MUC1* and does not bind to another form of cleaved MUC1 that is present on some normal tissues that also have a rapid turnover. To be clear, patients will receive either huMNC2-CAR44 or huMNC2-CAR22, but not a combined product.

The huMNC2-CAR44 product consists of autologous T cells that are isolated from cancer patients, transduced with a proprietary lentiviral vector backbone manufactured under cGMP and containing sequences for a human CD8 alpha leader sequence, humanized MNC2-scFv (MUC1* targeting head), portions of human CD8 hinge and transmembrane domains, and human 4-1BB and human CD3-zeta costimulatory domains. The huMNC2-CAR44 transduced T cells are antigen-stimulated in vitro, with a synthetic MUC1* extracellular domain peptide. The CAR T cells are then ready for administration to the patient. Alternatively, the CAR T cells can be cryopreserved, then administered to the patient after thaw at bedside.

The huMNC2-CAR22 product is comprised of a CD8-α leader sequence, the huMNC2 scFv, a CD28 hinge and transmembrane region, followed by a CD28 co-stimulatory domain and a CD3-ζ signaling domain bearing two Tyrosine to Phenylalanine mutations in each of ITAMs 2 and 3 to minimize CAR T cell exhaustion and increase in vivo persistence. The huMNC2-CAR22 transduced T cells are not antigen-stimulated. The CAR T cells can be cryopreserved, then administered to the patient after thaw at bedside.

The investigators propose to evaluate the safety and preliminary anti-tumor activity of adoptively transferred autologous T cells genetically modified to express a CAR that targets MUC1*, huMNC2-CAR44 or huMNC2-CAR22, in Phase I/II clinical trials in patients with metastatic MUC1* positive breast cancers.

ELIGIBILITY:
Please note that results of tests and/or procedures conducted as per standard of care purposes may be used for research purposes if conducted within the protocol-defined window prior to screening/leukapheresis and/or T-Cell Therapy.

Inclusion Criteria:

1. Confirmation of diagnosis of breast cancer by pathology review of initial or subsequent biopsy or other pathologic material at the City of Hope Pathology department. ER, PR, and HER2 status known and documented per ASCO/CAP guidelines.

   1. For dose expansion cohorts, tumors with ER and/or PR ≥1% will be considered hormone receptor positive. Tumors with ER and PR <1% will be considered hormone receptor negative. HER2 status will be determined by IHC or FISH per ASCO/CAP guidelines. Patients will be allocated to expansion cohorts according to guidelines in table below.
   2. Dose expansion cohorts

   Expansion Cohort Hormone Receptor status HER2 status Luminal ER and/or PR >/=1% positive Negative by IHC or FISH HER2 positive Any ER or PR status Positive by IHC or FISH Triple Negative ER and PR <1% Negative by IHC or FISH
2. Patients must have received standard metastatic systemic therapy per NCCN guidelines or institutional practice which are known to confer benefit. No maximum on number of prior systemic treatment regimens.

   1. Patients with hormone receptor positive disease must have received at least 3 prior endocrine therapies and at least 2 prior lines of chemotherapy in the metastatic setting.
   2. Patients with HER2 positive breast cancer must have received at least 3 prior HER2- directed therapies (trastuzumab, pertuzumab, TDM-1 or others) in the metastatic setting.
   3. Patients with triple negative disease must have received at least 2 prior lines of chemotherapy in the metastatic setting.
3. MUC1* membrane expression ≥30% by immunohistochemistry on a tumor specimen obtained at screening or previous tumor specimen that is less than 6-months old (see Appendix I for examples of MUC1* expression patterns).
4. Patients must be 18 years of age or older, of any gender, race or ethnicity.
5. Patients must be capable of understanding and providing a written informed consent.
6. Patients must have a Karnofsky performance status of ≥60%.
7. Patients must have measurable disease by at least one of the criteria below:

   1. Extra skeletal disease that can be accurately measured by CT or MRI per RECIST 1.1,
   2. Skeletal or bone-only metastases measurable by FDG PET imaging.
8. Negative serum pregnancy test within 14 days of planned leukapheresis and within 28 days of lymphodepleting chemotherapy for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year.
9. Fertile male and female patients must be willing to use an effective contraceptive method before, during, and for at least 4 months after the huMNC2-CAR T cell infusion.

Exclusion Criteria:

1. Patients requiring ongoing daily corticosteroid therapy at a dose of >15 mg of prednisone per day (or equivalent). Pulsed corticosteroid use for disease control is acceptable.
2. Active autoimmune disease requiring immunosuppressive therapy is excluded unless discussed with the PI.
3. Major organ dysfunction defined as:

   1. Serum creatinine > 2 mg/dL
   2. Bilirubin ≥ 1.5 mg/dL with the following exception: Patients with known Gilbert disease, serum bilirubin > 3 mg/dL
   3. AST or ALT ≥ 2.5 x upper institutional limit of normal with the following exception: Patients with known hepatic metastases, AST or ALT > 3x upper institutional limit of normal
   4. Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing. Those with an FEV1 of < 50 % of predicted or DLCO (corrected) < 40% will be excluded.
   5. Significant cardiovascular abnormalities as defined by any one of the following:

   i. NYHA class III or IV congestive heart failure, ii. clinically significant hypotension, iii. uncontrolled symptomatic coronary artery disease, or iv. a documented ejection fraction of <45%. Any patient with an EF of 45-49% must receive clearance by a cardiologist to be eligible for the trial.
4. ANC <1000/mm^3.
5. Hemoglobin <9 mg/dl (transfusion permitted to achieve this).
6. Platelet count <75,000/mm^3.
7. Treatment with investigational agent(s) within 30 days of planned lymphodepletion.
8. HIV seropositive.
9. Uncontrolled active infection.
10. Anticipated survival of <3 months.
11. Breast-feeding women.
12. Patients who have a contraindication to cyclophosphamide chemotherapy.
13. Known second malignancy that is progressing or requires active treatment.
14. Untreated CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate with documented stable disease as defined by no evidence of progression by imaging or symptoms for at least 4 weeks prior to enrollment.
15. Have psychiatric illness, social situation, or other medical condition that would preclude informed consent to limit compliance with study requirements, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2035-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Within 35 days after T cell infusion
  To determine the safety and maximally tolerated cell dose (MTD) and recommended phase 2 cell dose (RP2D) of ex vivo expanded autologous huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells for patients with advanced MUC1* positive breast cancer using CTCAE version 5.0 and Lee criteria.

SECONDARY OUTCOMES:
In vivo persistence | Up to 365 days after the T cell infusion
  Determine duration of in vivo persistence and phenotype of adoptively transferred huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells.
Preliminary Antitumor Activity | Up to 15 years
  Preliminary antitumor activity of the adoptive transfer of huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells in all patients with measurable tumor prior to T cell transfer by RECIST 1.1
Antitumor Activity | Up to 15 years
  Determine antitumor activity at MTD/RP2D of huMNC2-CAR44 T cells or huMNC2-CAR22 CAR T cells in patients with luminal breast cancer (hormone receptor positive, HER2 negative), HER2 positive breast cancer, and triple negative breast cancer (hormone receptor and HER2 negative) by RECIST 1.1 in expansion cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562